CLINICAL TRIAL: NCT00950768
Title: GISMM2001: Melphalan 200 mg/m2 Versus Melphalan 100 mg/m2 in Newly Diagnosed Myeloma Patients: a Prospective, Multi-center Phase III Study
Brief Title: Melphalan 200 mg/m2 Versus Melphalan 100 mg/m2 in Newly Diagnosed Myeloma Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda Ospedaliera San Giovanni Battista (Other)
Responsible Party: Mario Boccadoro, Division of Hematology - University of Torino - A.O.U. San Giovanni Battista
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GISMM2001
Record Dates: First submitted 2009-07-31; First posted 2009-08-03 (Estimated); Last update posted 2009-08-03 (Estimated); Status verified 2009-07

CONDITIONS: Multiple Myeloma; Diagnosis
Keywords: Myeloma; Melphalan; Autologous transplantation
MeSH Terms: conditions — Multiple Myeloma; Disease; Neoplasms, Plasma Cell | interventions — Transplantation, Autologous

ARMS (2):
- Mel100 (Active Comparator)
  Interventions: Procedure: Autologous transplantation
- Mel200 (Experimental)
  Interventions: Procedure: Autologous transplantation

INTERVENTIONS:
Procedure: Autologous transplantation — Tandem autologous transplantation Melphalan 100 mg/m2 versus Melphalan 200 mg/m2

SUMMARY:
In this study will be randomised before induction treatment either to receive two courses of melphalan 200 mg/m2 (MEL200) or two courses of melphalan 100 mg/m2 (MEL100). Informed consent will be obtained upon enrolment. Inclusion criteria included: diagnosis of untreated Durie e Salmon stage IIA-IIIB measurable multiple myeloma; age < 65 years. Exclusion criteria included: prior treatment for myeloma; abnormal cardiac function, defined as systolic ejection fraction <50%; abnormal pulmonary spirometry test; serum bilirubins > 2.5 times normal and ALAT and/or ASAT > 2 times normal; seropositivity for HIV, HCV or HBV, active non-hematologic malignancies.

Induction therapy, PBSC mobilization, and autografting Initial treatment plan included induction chemotherapy with 2 courses of vincristine, 1 mg/m2 on day 1, adriamycin, 50 mg/m2 on day 1, and dexamethasone, 40mg/day days 1-4, administered 28 days apart, followed by peripheral blood stem cell (PBSC) mobilisation and harvest after 1 or 2 cycles of cyclophosphamide, 4 g/m2, and G-CSF, 10 ug/kg given i.v. or subcutaneously. After at least one month from PBSC collection, autografting consisted of melphalan, 200 mg/m2 or melphalan, 100 mg/m2, on day -2, and cryopreserved PBSC infusion on day 0. Patients received G-CSF, 5 ug/kg, from days +3 until neutrophil count > 1000/ul were achieved.

Supportive care and toxicity grading Following autografting, all patients received standard prophylaxis against bacterial and fungal infections; herpes simplex and varicella-zoster virus reactivation; and Pneumocystis carinii. Cytomegalovirus CMV reactivation was monitored through levels of CMV antigenemia and/or serum CMV DNA levels and treated with ganciclovir or foscarnet as clinically indicated. Standard criteria (Common Toxicity Criteria version 3.0) were used for grading hematological and non-hematological toxicity.

ELIGIBILITY:
Inclusion criteria included:

* diagnosis of untreated Durie & Salmon stage IIA-IIIB measurable multiple myeloma;
* age < 65 years.

Exclusion criteria included:

* prior treatment for myeloma;
* abnormal cardiac function, defined as systolic ejection fraction <50%;
* abnormal pulmonary spirometry test;
* serum bilirubins > 2.5 times normal and ALAT and/or ASAT > 2 times normal;
* seropositivity for HIV, HCV or HBV, active non-hematologic malignancies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2002-02; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Primary endpoints of the study were Overall Survival defined as the time from diagnosis until death from any cause; Progression Free Survival defined as the time from diagnosis until death from any cause or date of first relapse or progression.

SECONDARY OUTCOMES:
Secondary endpoint was time to progression (TTP) defined as the time from the date of diagnosis to relapse or death from progression.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Boccadoro, MD, Principal Investigator — Division of Hematology - University of Torino - A.O.U. San Giovanni Battista

REFERENCES:
- [Derived] Palumbo A, Bringhen S, Bruno B, Falcone AP, Liberati AM, Grasso M, Ria R, Pisani F, Cangialosi C, Caravita T, Levi A, Meloni G, Nozza A, Pregno P, Gabbas A, Callea V, Rizzo M, Annino L, De Stefano V, Musto P, Baldi I, Cavallo F, Petrucci MT, Massaia M, Boccadoro M. Melphalan 200 mg/m(2) versus melphalan 100 mg/m(2) in newly diagnosed myeloma patients: a prospective, multicenter phase 3 study. Blood. 2010 Mar 11;115(10):1873-9. doi: 10.1182/blood-2009-09-241737. Epub 2009 Dec 1. PMID 19965659